CLINICAL TRIAL: NCT06368154
Title: Prospective Cohort Study of Exosomal microRNAs as Biomarkers for Diagnosis and Therapeutic Efficacy Evaluation of Metabolic Bone Diseases in Premature Infants
Brief Title: Exosome microRNAs as Potential Biomarkers of Metabolic Bone Disease of Prematurity
Status: Recruiting | Type: Observational
Sponsor: Hunan Children's Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: HCHLL-2019-08
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2023-11

CONDITIONS: Exosomes; Newborn; Bone Diseases, Metabolic
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Less than 32 weeks: The gestational age was less than 32 weeks, there was no history of surgery, blood transfusion, congenital malformation and inherited metabolic diseases. The corrected gestational age of less than 44 weeks。
- 32 to 36+6 weeks: The gestational age was 32-36+6 weeks, there was no history of surgery, blood transfusion, congenital malformation and inherited metabolic diseases. The corrected gestational age of less than 44 weeks。
- control group: Term infants with a gestational age of 37+0-41+6 weeks, no blood transfusion, no surgery, no congenital malformation, no inherited metabolic diseases, no history of parenteral nutrition, no intestinal diseases. The corrected gestational age of less than 44 weeks.

SUMMARY:
Metabolic bone disease of prematurity (MBDP) is caused by insufficient content of calcium, phosphorus, and organic protein matrix in preterm infants or bone metabolism disorder, which is one of the complications affecting the quality of life of preterm infants. The early symptoms of MBDP are insidious, and there is no unified and clear diagnostic method. The diagnosis is mostly based on typical clinical manifestations and X-ray findings, but at this time, bone mineral density has decreased significantly, so early detection and diagnosis are difficult. Studies have shown that exosomal micrornas have biological characteristics and targeting specificity, and can be used as new molecular diagnostic markers for diseases. Several studies have reported the use of plasma or serum microRNAs as molecular markers for early prediction of bone diseases. In our previous study, we extracted plasma exosomes from preterm infants for high-throughput sequencing of microRNAs, and identified differentially expressed micrornas related to bone metabolism. In this study, exosomes were used as carriers, and digital PCR was used to verify the specificity and sensitivity of plasma exosomal microRNA as biomarkers of MBDP in a large sample size. The above biomarkers were compared and verified before and after treatment in children with MBDP. Further revealing plasma exosomal microRNA as a biological indicator for evaluating the efficacy of MBDP may improve the diagnostic level of MBDP, improve the outcome and prognosis of very low birth weight preterm infants, thereby improving global health and reducing socioeconomic costs.

ELIGIBILITY:
Inclusion Criteria:

* The gestational age was 37+0-41+6 weeks and the age was less than 28 days

Exclusion Criteria:

* There was no blood transfusion, no operation, no congenital malformation, no inherited metabolic diseases, no history of intravenous nutrition, and no intestinal diseases

Ages: 0 Hours to 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Gestational age < 37 weeks, corrected gestational age < 44 weeks, there was no history of surgery, blood transfusion, congenital malformation and inherited metabolic diseases.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
exosomes | 6 months of age
  Plasma exosomal digital PCR was used for microRNA validation

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Children's Hospital, Changsha, Hunan, China